CLINICAL TRIAL: NCT04686123
Title: Effectiveness of Strengthening and Stretching Exercise on the Resting Length of Pectoralis Minor Muscle and Shoulder Flexion of Young Females With Rounded Shoulder Posture
Brief Title: Efficacy of a Supervised Intervention Protocol on Rounded Shoulder Posture and Shoulder ROM Among Saudi Young Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Majmaah University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-21
Record Dates: First submitted 2020-12-24; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Postural; Defect
Keywords: Round shoulder posture; Active Stretching; Pectoralis Muscles; Strength Training; Trapezius Muscle
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Two-arm parallel groups randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A performed active Stretching of Pectoralis Minor (PMi) muscle along with the strengthening of Lower Trapezius muscle under the supervision of a physiotherapist
  Interventions: Other: Active Stretching or Self-stretching exercises; Other: Active strengthening Or Self-Strengthening exercises
- Group B (Active Comparator): Group B performed active Stretching of the Pectoralis Minor (PMi) muscle only under the supervision of a physiotherapist.
  Interventions: Other: Active Stretching or Self-stretching exercises

INTERVENTIONS:
Other: Active Stretching or Self-stretching exercises — Pectoralis minor muscle was actively stretched under the supervision of a physiotherapist as follows: - 2 sets of 3-stretches/session/day, for 5 consecutive days a week, for 3 weeks
Other: Active strengthening Or Self-Strengthening exercises — Lower trapezius muscle was strengthened under the supervision of a physiotherapist as follows: -2 sets of 5-rep./session/day, for 5 consecutive days in 1st week, progressed to 10 and 20 reps./session/day for 2 weeks and 3 weeks respectively.
  Arms: Group A

SUMMARY:
Shortening of pectoralis minor (PMi) muscle affects the scapular excursion that results in limited shoulder flexion range of motion (SFROM). The purpose is to evaluate the effect of Stretching of PM muscle along with the strengthening of lower trapezius (LTR) muscle to increase the length of PM muscle (PML) and limited SFROM in young adult females with rounded shoulder posture.

DETAILED DESCRIPTION:
Shortening of pectoralis minor (PMi) muscle affects the scapular excursion that results in limited shoulder flexion range of motion (SFROM). The purpose is to evaluate the effect of Stretching of PM muscle along with the strengthening of lower trapezius (LTR) muscle to increase the length of PM muscle (PML) and limited SFROM in young adult females with rounded shoulder posture.

Randomized sixty female subjects with rounded shoulder posture into two groups: Group A performed active Stretching of PMi along with the strengthening of LTR muscle(n=30); group B performed dynamic Stretching of PMi muscle only. Scores of outcome measures were recorded before and post interventions on day 0, day10th, and day21st, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Young Adult Female having a PMLD test score of more than 2.5cm
* Aged between 20-30 years
* No history of shoulder trauma or current shoulder pathology, thoracic scoliosis, or kyphosis deformity.
* Showed self-cooperation for the study

Exclusion Criteria:

* Young Adult Female having a PMLD test score of equal to or less than 2.5cm
* History of shoulder trauma or current shoulder pathology, thoracic scoliosis, or kyphosis deformity.
* Showed non-cooperation for the study

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity.
Enrollment: 60 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Resting length of Pectoralis Minor (PMi) muscle | 3-weeks
  It was assessed by Pectoralis Minor Length Distance Test (PMLDT)
Shoulder Flexion Range of Motion (SFROM) | 3-weeks
  It was assessed by a Universal Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT-Ortho, Principal Investigator — King Saud University
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No